CLINICAL TRIAL: NCT01578135
Title: French National Longitudinal Prospective Follow-up of Children Born Small for Gestational Age and Treated With Norditropin SimpleXx (French Health Authorities Commitment)
Brief Title: French National Registry of Children Born Small for Gestational Age Treated With Somatropin
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GHSGA-1757
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Growth Disorder; Small for Gestational Age
MeSH Terms: conditions — Growth Disorders | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase I
  Interventions: Drug: somatropin
- Phase II
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Patients are to fill in a questionnaire at inclusion in registry
  Groups: Phase I
Drug: somatropin — Patients are to fill in a questionnaire 6 months after inclusion into registry and then annually until adult height is reached
  Groups: Phase II

SUMMARY:
This study is conducted in Europe. The aim of the study is to describe the patient population and therapeutic practices (study phase I), assess efficacy on growth and adult height and assess tolerance of somatropin (Norditropin® SimpleXx®) (study phase II)

ELIGIBILITY:
Inclusion Criteria:

* Born small for gestational age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Phase I: All patients born SGA treated with Norditropin® SimpleXx® (somatropin) whether they were previously treated with another growth hormone for this indication or not from the 29th of April 2005 until 29th of April 2010.
  Phase II: Sub-population randomly selected (every 5th patient being included in registry in study phase I).
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2007-03-18 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Growth in height | 6 months after inclusion into registry and then annually until adult height is reached

SECONDARY OUTCOMES:
Blood pressure: Systolic and diastolic | 6 months after inclusion into registry and then annually until adult height is reached
Bone age | 6 months after inclusion into registry and then annually until adult height is reached
Insulin-Like Growth Factor 1 (IGF-1) | 6 months after inclusion into registry and then annually until adult height is reached

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Paris La Défense, France

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com